CLINICAL TRIAL: NCT02872844
Title: Local Heat-Stress as a Mechanism of Hearing Preservation in Adults Treated With Cisplatin: A Pilot Study
Brief Title: Local Heat-Stress as a Mechanism of Hearing Preservation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator closed study-no accrual
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0170-16-FB
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Heat-stress (Experimental): Each participant will undergo a 30-minute heat stress to one randomized ear. The participant will be reclined and the hot air caloric at 50°C applied by a licensed, unblinded audiologist for 30 minutes.
  Interventions: Device: ICS AirCal3

INTERVENTIONS:
Device: ICS AirCal3 — Each patient will undergo a 30-minute heat stress to one ear. For randomization, the left ear will be treated in patients with a registration number ending with an odd number and the right for even numbers. An ICS AirCal3 Research Strategy (Otometrics) system attached to an Intel Core 15vPro Thinkpad (IBM) laptop is used within the audiometry department of a separate outpatient clinic. The patients will be reclined and the hot air caloric at 50°C applied by a licensed, unblinded audiologist for 30 minutes. The patients will be allowed to fixate and use whatever means they prefer for entertainment during the intervention.

SUMMARY:
This pilot study plans to determine whether or not local heat-stress as a mechanism can help to preserve hearing in adults treated with Cisplatin.

DETAILED DESCRIPTION:
Evidence from the laboratory over the past 10-15 years has demonstrated that heat stress to the ear is otoprotectant against a variety of insults. The strongest evidence supports heat-shock protein 70 (Hsp70) as a key facilitator in this protection. Hsp70 is well established as a cell stabilizer, especially for cells undergoing significant stress. Hsp70 has been shown to protect against cisplatin-induced ototoxicity. Induction of Hsp70 may be accomplished pharmacologically, by whole-body heat stress, or by local heat stress. A form of local heat-stress is already employed in the common clinical setting of the warm caloric. This vestibular test has been in place since the early 20th century with a variety of studies evaluating the patient vestibular response to a variety of times and temperatures. Current clinical practice recommends either water or air calorics of 45°C or 50°C (respectively) at 45-60 seconds.

Several studies have described administering prolonged caloric stimulation to individual subjects without ill effect. Patients are able to tolerate stimulation up to 60 minutes without intolerable nystagmus or vertiginous symptoms or significant injury. Thus, it is feasible to provide warm stimulus to the ear for the recommended time of 30 minutes at the recommended temperature of 50°C (air) without significant risk to the patient.

The purpose of this study is to evaluate the impact of heat stress to the inner ear as an otoprotectant intervention against cisplatin-induced hearing loss. Patients that meet inclusion criteria will be offered audiometric evaluation before each cisplatin treatment and at 1, 3, 6, and 12 months following their chemotherapy. Patients will undergo their heat-stress 5-7 hours prior to their cisplatin treatment. Patients will serve as their own controls with one ear randomly receiving treatment and the other not. The primary outcome will be audiometric testing. Blood samples will be collected for serum levels of Hsp70 as a secondary outcome. A sample size of 12 achieves 80% power to detect a 0.9 standard deviation difference between ears using a two-sided paired t-test at 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing total cisplatin in total doses > 100mg/m2.
* Written consent.
* Age > 19 years.

Exclusion Criteria:

* Inability to tolerate the intervention
* Exposure to cisplatin treatment without intervention.
* Head and neck carcinoma
* Baseline asymmetric hearing loss.
* Pregnant or breastfeeding women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Audiometric Effect | One year
  Audiometric evaluation will serve as the primary measure of outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Judge, MD, Principal Investigator — University of Nebraska